CLINICAL TRIAL: NCT03922347
Title: Modelling and Evaluation of a Community-oriented mHealth-based Screening and Promotional Programme for Improving Eye Health in Iran
Brief Title: mHealth Intervention for Improving Eye Health at Community Level
Acronym: Vison mHealth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Head of ophthalmic research center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 96315
Record Dates: First submitted 2019-04-13; First posted 2019-04-19 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Visual Impairment
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- routine care (No Intervention)
- Screening program including 2 consecutive tests (Active Comparator)
  Interventions: Diagnostic Test: Screening program including 2 consecutive tests
- Screening program with mobile health (Active Comparator)
  Interventions: Diagnostic Test: Screening program with mobile health

INTERVENTIONS:
Diagnostic Test: Screening program including 2 consecutive tests — visual acuity test by Snellen chart, fundus imaging by fundus photography (Visucam Pro NM; Carl Zeiss Meditec AG, Germany)
  Arms: Screening program including 2 consecutive tests
Diagnostic Test: Screening program with mobile health — Peek Acuity and Peek Retina installed on smart phones (Samsung Galaxy S8)
  Arms: Screening program with mobile health

SUMMARY:
This study is a community trial that aims to establish and evaluate an mHealth screening and promotional tool for improving eye health in Iran. Sampling frame is a region in Tehran province with around 1 million sub-urban and rural inhabitants. investigators have obtained the list of health centers and their underserved population from the health authorities. In this region, health services are delivered through rural health houses, urban health posts and overhead health centers (221 units in total). investigators choose 27 units using cluster random sampling method with a probability proportional to size strategy, then investigators randomly assign them into three arms (explained below). The interventions will be at community level with the community as the unit of randomization.

Arm 1- Training of the Primary Health Care (PHC) workers + PHC workers will be empowered with the mHealth tool to monitor, screen and promote community members Arm 2- PHC system will be strengthened with health promotion and screening programmes (same content as the mHealth tool) and PHC workers will deliver eye health messages and screening tests by the conventional facilities.

Arm 3: Control group: only observation and registering of routine care

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were living in one of the non-institutionalized urban or rural residential areas in one of the survey area, being resident in the same address for at least 6 months during the year before the enrolment, age 50 and over and Iranian nationality.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3300 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Eye care utilization: being visited/treated by an eye care professional | 6-12 months
  Questionnaire based on closed questions

SECONDARY OUTCOMES:
Visual acuity | At baseline
  Peek Acuity Software installed on smart phones (Samsung Galaxy S8, based on Logarithm Minimum Angle of Resolution, LogMAR). Visual acuity will be presented in range (minimum to maximum).
  Higher value of visual acuity represents the worsened outcome.
fundus imaging | At baseline
  Peek Retina Software installed on smart phones (Samsung Galaxy S8; based on Logarithm Minimum Angle of Resolution, LogMAR). Higher value of visual acuity represents the worsened outcome.
Based on Logarithm Minimum Angle of Resolution, LogMAR. Visual acuity will be presented in range (minimum to maximum). Higher value of visual acuity represents the worsened outcome. | At baseline
  visual acuity test by Snellen chart
fundus imaging by fundus photography (Visucam Pro NM; Carl Zeiss Meditec AG, Germany) | At baseline
  fundus photography (Visucam Pro NM; Carl Zeiss Meditec AG, Germany)

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Iran